CLINICAL TRIAL: NCT00736177
Title: Comparison of Transfers of Fresh and Thawed Embryos in Patients With Prior Failed Embryo Transfer Cycles
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment
Sponsor: Fertility Center of Las Vegas (Industry)
Responsible Party: Bruce Shapiro, M.D., Medical Director, Fertility Center of Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAIRB-08-0012
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2009-02

CONDITIONS: Infertility; Subfertility
Keywords: IVF; blastocyst transfer; endometrium; embryo cryopreservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients in the control group will undergo conventional IVF cycles with fresh blastocyst transfer.
  Interventions: Procedure: Fresh embryo transfer
- Test group (Experimental): Patients in the Test group will have their embryos cryopreserved for transfer in a second cycle.
  Interventions: Procedure: Embryo cryopreservation

INTERVENTIONS:
Procedure: Embryo cryopreservation — Subjects in the Test group will have their embryos cryopreserved for transfer in a subsequent cycle.
  Arms: Test group
Procedure: Fresh embryo transfer — Subjects in the Control group will receive fresh embryo transfer.
  Arms: Control

SUMMARY:
This study seeks to determine if patients with a history of failed fresh embryo transfer(s) will have increased success rates with embryo cryopreservation and subsequent thawed embryo transfer when compared to fresh embryo transfer.

DETAILED DESCRIPTION:
Implantation failure remains a significant problem in cycles of in vitro fertilization (IVF). Patients with a history of implantation failure in fresh autologous cycles have been shown have reduced chance of success in subsequent fresh autologous cycles. A potentially frequent cause of implantation failure is reduced endometrial receptivity following ovarian stimulation, perhaps due to the effects of supraphysiologic hormone levels on endometrial development. Therefore, such patients may have a greater chance of success if all of their embryos are cryopreserved for use in a subsequent cycle in which endometrial development can be more carefully controlled, absent the effects of ovarian stimulation. Therefore this study compares success rates in cycles of fresh embryo transfer and cycles with transfer of frozen-thawed embryos.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* Cycle day 3 FSH less than 10 IU/l
* At least 8 antral follicles
* At least one previous autologous embryo transfer cycle that did not result in ongoing pregnancy at 10 weeks.

Exclusion Criteria:

* Embryo biopsy
* Any prior fresh embryo transfer that resulted in live birth

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy with fetal heart motion | 10 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shapiro, M.D., Principal Investigator — Fertility Center of Las Vegas
Locations (1):
- Fertility Center of Las Vegas, Las Vegas, Nevada, United States

REFERENCES:
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Thomas S. Large blastocyst diameter, early blastulation, and low preovulatory serum progesterone are dominant predictors of clinical pregnancy in fresh autologous cycles. Fertil Steril. 2008 Aug;90(2):302-9. doi: 10.1016/j.fertnstert.2007.06.062. Epub 2007 Oct 1. PMID 17905239
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Ross R. Contrasting patterns in in vitro fertilization pregnancy rates among fresh autologous, fresh oocyte donor, and cryopreserved cycles with the use of day 5 or day 6 blastocysts may reflect differences in embryo-endometrium synchrony. Fertil Steril. 2008 Jan;89(1):20-6. doi: 10.1016/j.fertnstert.2006.08.092. Epub 2007 Jan 16. PMID 17224151
- See also: Fertility Center of Las Vegas — http://www.fertilitycenterlv.com